CLINICAL TRIAL: NCT03613324
Title: Prevalence Rates of Bladder Outlet Obstruction and Detrusor Underactivity and Their Clinical and Urodynamic Findings in Women With ≥Stage II Cystocele
Brief Title: BOO and DU and Their Clinical and Urodynamic Findings in Women With ≥Stage II Cystocele
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805025RINB
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Bladder Outlet Obstruction and Detrusor Underactivity in Women With Severe Cystocele
Keywords: Cystocele; Bladder outlet obstruction; Detrusor underactivity; Urodynamic study
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Cystocele; Urinary Bladder, Underactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bladder outlet obstruction (BOO): Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20 min pad testing and urodynamic studies in a medical center were reviewed. Woman were defined as having BOO when Qmax was <12 mL/s and PdetQmax was ≥25 cmH2O with sustained detrusor contraction during voiding cystometry.
  Interventions: Diagnostic Test: Pad test
- Detrusor underactivity (DU): Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20 min pad testing and urodynamic studies in a medical center were reviewed. Woman were defined as having DU when Qmax was <12 mL/s and PdetQmax was <10 cmH2O during voiding cystometry.
  Interventions: Diagnostic Test: Pad test
- ND BOO/DU: Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20 min pad testing and urodynamic studies in a medical center were reviewed. This group revealed no demonstrated bladder outlet obstruction nor detrusor underactivity.
  Interventions: Diagnostic Test: Pad test

INTERVENTIONS:
Diagnostic Test: Pad test — 20-minutes pad test and urodynamic study including uroflowmetry, filling cystometry and voiding cystometry.
  Other Names: Urodynamic study

SUMMARY:
Prevalence rates of bladder outlet obstruction (BOO) and detrusor underactivity (DU) and their related clinical and urodynamic findings in women with ≥ pelvic organ prolapse quantification stage II cystocele are important for clinical consultation. Thus, the aim of this study was to elucidate the above findings and between-group associations.

DETAILED DESCRIPTION:
Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20 min pad testing and urodynamic studies in a medical center were reviewed. Only those with complete data of maximum flow rate (Qmax) and detrusor pressure at maximum flow rate (PdetQmax) were enrolled. ANOVA test and post-hoc testing with bonferroni's correction were used for statistical analysis. Woman were defined as having DU when Qmax was <12 mL/s and PdetQmax was <10 cmH2O, and were defined as having BOO when Qmax was <12 mL/s and PdetQmax was ≥25 cmH2O with sustained detrusor contraction during voiding cystometry.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20y/o
2. Cystocele > stage II
3. Complete pad test and urodynamic study

Exclusion Criteria:

1. Pregnancy
2. Urinary tract infection
3. Had received pelvic reconstruction surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with more than stage II cystocele
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
BOO | November 2011 to January 2017
  Bladder outlet obstruction: Qmax was <12 mL/s and PdetQmax was ≥25 cmH2O with sustained detrusor contraction during voiding cystometry.
DU | November 2011 to January 2017
  Detrusor underactivity: <12 mL/s and PdetQmax was <10 cmH2O

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD